CLINICAL TRIAL: NCT00435929
Title: Effect of Moderate Liver Impairment on the Pharmacokinetics of Saquinavir After Administration of Saquinavir/Ritonavir 1000/100mg BID in HIV Patients
Brief Title: A Study of Saquinavir/Ritonavir in Liver-Impaired Patients With HIV Infection.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP17921
Record Dates: First submitted 2007-02-15; First posted 2007-02-16 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-02

CONDITIONS: HIV Infections
Keywords: Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir; Saquinavir

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Ritonavir; Drug: saquinavir [Invirase]
- 2 (Experimental)
  Interventions: Drug: Ritonavir; Drug: saquinavir [Invirase]

INTERVENTIONS:
Drug: Ritonavir — 100mg po bid
Drug: saquinavir [Invirase] — 1000mg po bid

SUMMARY:
This 2 arm study will assess the effect of moderate liver impairment on the pharmacokinetics of saquinavir and ritonavir at steady state following administration of saquinavir/ritonavir 1000mg/100mg po bid in HIV patients. Saquinavir/ritonavir will be administered concomitantly with 2 to 3 active nucleoside reverse transcriptase inhibitors. The study will compare a group of HIV patients without known liver disease and a group with moderate liver disease. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* HIV infection;
* normal liver function, or moderate liver disease (Child-Pugh grade B);
* antiretroviral therapy naive and eligible to take antiretroviral treatment as per treatment guidelines, or treatment experienced for at least 4 weeks prior to first dosing.

Exclusion Criteria:

* severe ascites at screening, or Child-Pugh grade C;
* acute infection or current malignancy requiring treatment;
* taking any inhibitor of CYP3A4 (with the exception of anti-HIV drugs) within 14 days prior to first dosing;
* taking any inducer of CYP3A4 (with the exception of anti-HIV drugs) within 4 weeks prior to pharmacokinetic evaluation (day 14 or 28);
* evidence of resistance to saquinavir.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-09; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (8):
- United States (5):
  - Chicago, Illinois
  - Somers Point, New Jersey
  - Voorhees Township, New Jersey
  - Philadelphia, Pennsylvania
  - Dallas, Texas
- Canada (2):
  - Ottawa, Ontario
  - Toronto, Ontario
- San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 12 September 2006 to 09 April 2009 at 3 sites in US and 2 in Canada.
Pre-assignment Details: Total 19 participants were screened. A total 9 participants with HIV infection with moderate liver disease (Group 2) and 7 participants with HIV infection with normal liver function (Group 1) were enrolled in the study. Participants in Group 1 were matched with those in Group 2 on the basis of age, gender, weight, and tobacco use.
Groups:
- Normal Liver Function: Participants with human immunodeficiency virus (HIV) infection and with normal liver function receiving saquinavir (SQV)/ritonavir (RTV) 1000/100 mg orally twice a day (BID) for 14 days.
- Moderate Hepatic Impairment: Participants with HIV infection and with moderate hepatic impairment receiving SQV/RTV 1000/100 mg orally BID for 14 days.
Period: Overall Study
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 9 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time of Administration to 12 Hours After Dosing (AUC 0-12h) of Saquinavir (SQV) and Ritonavir (RTV)
Description: Area Under the Plasma Concentration-Time Curve (AUC) is a measure of the plasma concentration of the drug over time. It is used to characterize drug absorption. The pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the area under the plasma concentration-time curve from 0 to 12 hours after dosing (AUC (0-12h) of SQV and RTV The AUC (0-12hours) was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post-dose on Day 14
Population: Pharmacokinetic (PK) analysis population: All participants who adhered to the study protocol and had evaluable concentration data and PK parameters on Day 14.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
ng*hr/mL
  AUC for SQV | 28518 (20157) | 24332 (24700)
  AUC for RTV | 10985 (1723) | 9930 (5243)
Statistical Analysis 1: Comparison: Normal Liver Function vs Moderate Hepatic Impairment; Comparison between normal liver function and moderate hepatic impairment for SQV; Test type: Superiority or Other; Geometric mean ratio = 0.656, 90% CI 2-sided [0.268 to 1.603]
Statistical Analysis 2: Comparison: Normal Liver Function vs Moderate Hepatic Impairment; Comparison between normal liver function and moderate hepatic impairment for RTV; Test type: Superiority or Other; Geometric mean ratio = 0.764, 90% CI 2-sided [0.505 to 1.156]

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of SQV and RTV
Description: The plasma concentration (Cmax) is defined as maximum observed analyte concentration. The pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the maximum observed plasma concentration (C max) of SQV and Ritonavir RTV The Cmax was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post-dose on Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
ng/mL
  Cmax of SQV | 4300 (2940) | 3610 (3000)
  Cmax of RTV | 1500 (294) | 1460 (690)
Statistical Analysis 1: Comparison: Normal Liver Function vs Moderate Hepatic Impairment; Comparison between normal liver function and moderate hepatic impairment for SQV; Test type: Superiority or Other; Geometric Mean Ratio = 0.716, 90% CI 2-sided [0.311 to 1.644]
Statistical Analysis 2: Comparison: Normal Liver Function vs Moderate Hepatic Impairment; Comparison between normal liver function and moderate hepatic impairment for RTV; Test type: Superiority or Other; Geometric mean ratio = 0.844, 90% CI 2-sided [0.551 to 1.292]

3. Secondary Outcome: Time of Maximum Plasma Concentration (Tmax) of SQV and RTV
Description: The Tmax is defined as actual sampling time to reach maximum observed analyte concentration. The Pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the time of maximum plasma concentration of SQV and RTV. The Tmax was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post-dose on Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
hour
  Tmax of SQV | 5.00 (1.83) | 5.00 (2.38)
  Tmax of RTV | 4.29 (1.50) | 4.07 (1.75)

4. Secondary Outcome: Terminal Half-life (T1/2) of SQV and RTV
Description: Terminal half-life is the time measured for the plasma concentration to decrease by one half. The Pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the terminal half-life (T1/2) of SQV and RTV. The T1/2 was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post-dose on Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
hour
  T1/2 of SQV | 3.31 (0.823) | 4.10 (1.90)
  T1/2 of RTV | 3.80 (0.908) | 4.82 (2.82)

5. Secondary Outcome: Minimum Observed Plasma Concentration (Cmin) of SQV and RTV
Description: Cmin is the minimum blood plasma concentration that a drug achieves. The Pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the minimum observed plasma concentration (C min) of SQV and RTV The Cmin was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post dose on Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
ng/mL
  Cmin of SQV | 965 (920) | 834 (870)
  Cmin of RTV | 399 (172) | 418 (300)

6. Secondary Outcome: Plasma Clearance After Oral Administration (CL/F) of SQV and RTV
Description: The CL/F is the oral clearance; that is clearance based on oral bioavailability. The Pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the plasma clearance after oral administration (CL/F)of SQV and RTV The CL/F was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post dose on Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
L/hr
  CL/F of SQV | 47.052 (20.254) | 84.416 (68.645)
  CL/F of RTV | 9.289 (1.392) | 12.568 (5.885)

7. Secondary Outcome: Volume of Distribution (Vd) of SQV and RTV
Description: Vd is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. The pharmacokinetic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the Vd of SQV and RTV The Vd was analyzed for SQV and RTV by non-compartmental methods, using WinNonlin.
Time Frame: Pre-dose and at 0.5 hr, 1hr, 2hrs, 3hrs, 4hrs, 5hrs, 6hrs, 8hrs, 10hrs, and 12 hrs post dose on Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Litres
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
Litres
  Vd of SQV | 213.294 (95.048) | 464.049 (334.460)
  Vd of RTV | 50.232 (11.888) | 102.585 (112.579)

8. Secondary Outcome: Cluster of Differentiation 4 (CD4 ) Count
Description: The pharmacodynamic profile for following 14 days of administration with SQV/RTV 1000/100 mg BID included determining the cluster of differentiation 4 (CD4) count in participants in each group.
Time Frame: Screening (Day -35 to -1), pre-dose on Day 8, Day 14 and at follow up (Day 28-Day 35)
Population: PD analysis population: All participants who received at least 1 dose of the study medication and had at least 1 pharmacodynamic (PD) measure were included in the PD analysis population.
Measure: Mean (Standard Deviation); unit: cells/cubic millimeter
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 7
cells/cubic millimeter
  Screening; n=7, 9 | 540.000 (218.187) | 451.444 (249.011)
  Day 8;n=6, 9 | 638.500 (254.358) | 558.000 (243.994)
  Day 14;n=7, 9 | 683.571 (250.160) | 566.333 (257.484)
  Follow up; n=6, 8 | 692.500 (150.045) | 567.625 (261.947)

9. Secondary Outcome: Number of Participants With the Indicated Grade 3 and Grade 4 Laboratory Parameters
Description: Laboratory parameters specified in Clinical Operating Guidelines (COG) were summarized. AIDS Clinical Trial Group (ACTG) and American Heart Association (AHA) criteria were used to grade COG laboratory test values. Laboratory parameters for which an increase to Grade 3 (G3) or Grade 4 (G4) occurred are presented in the table below.
Time Frame: Up to Day 35
Population: Safety population: All participants who received at least 1 dose of study medication (whether or not they were withdrawn prematurely) and had safety follow-up data were included in safety analysis.
Measure: Number; unit: participants
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 9
participants
  ASAT (SGOT), (Hyper) G3 | 0 | 1
  ASAT (SGOT), (Hyper) G4 | 0 | 0
  Alkaline Phosphatase, (Hyper) G3 | 0 | 0
  Alkaline Phosphatase, (Hyper) G4 | 0 | 0
  ALAT (SGPT), (Hyper) G3 | 0 | 0
  ALAT (SGPT), (Hyper) G4 | 0 | 0
  Direct Bilirubin, (Hyper) G3 | 0 | 1
  Direct Bilirubin, (Hyper) G4 | 0 | 1
  Creatinine, (Hyper) G3 | 0 | 0
  Creatinine, (Hyper) G4 | 0 | 0
  Albumin, (Hypo) G3 | 0 | 0
  Albumin, (Hypo) G4 | 0 | 0
  Prothrombin Time seconds(Hyper) G3 | 0 | 1
  Prothrombin Time seconds (Hyper) G4 | 0 | 0
  Creatine Kinase, (Hyper) G3 | 0 | 1
  Creatine Kinase, (Hyper) G4 | 0 | 0
  Cholesterol, (Hyper) G3 | 0 | 0
  Cholesterol, (Hyper) G4 | 0 | 0
  Triglycerides, (Hyper) G3 | 2 | 0
  Triglycerides, (Hyper) G4 | 0 | 0
  Calcium, (Hypo) G3 | 0 | 0
  Calcium, (Hypo) G4 | 0 | 0
  Potassium, (Hypo) G3 | 0 | 0
  Potassium, (Hypo) G4 | 0 | 0
  Sodium, (Hypo) G3 | 0 | 0
  Sodium, (Hypo) G4 | 0 | 0
  Platelets, (Hypo) G3 | 0 | 0
  Platelets, (Hypo) G4 | 0 | 0
  Neutrophils, (Hypo) G3 | 0 | 1
  Neutrophils, (Hypo) G4 | 0 | 0
  Fasting Glucose, (Hyper) G3 | 0 | 0
  Fasting Glucose, (Hyper) G4 | 0 | 0
  Amylase, (Hyper) G3 | 0 | 1
  Amylase, (Hyper) G4 | 0 | 0
  Uric Acid, (Hyper) G3 | 0 | 2
  Uric Acid, (Hyper) G4 | 0 | 0
  Proteinuria 0 to 4+, (Hyper) G3 | 0 | 1
  Proteinuria 0 to 4+, (Hyper) G4 | 0 | 0

10. Secondary Outcome: Number Participants With Abnormal Vital Signs
Description: Abnormal Vital signs included are high and low Pulse rate (PR), high and how Temperature (Temp), high and low Systolic Blood Pressure (SBP) and high and low Diastolic Blood Pressure (DBP). Vital signs (SBP, DBP, PR,Temp) were measured after participants were in a semi-supine position for at least 5 minutes.
Time Frame: Up to Day 35
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 9
participants
  High PR | 0 | 0
  Low PR | 0 | 0
  High Temp | 0 | 0
  Low Temp | 0 | 0
  High-SBP | 1 | 1
  Low-SBP | 0 | 0
  High-DBP | 0 | 0
  Low-DBP | 1 | 2

11. Secondary Outcome: Number of Participants With Abnormal Electrocardiogram (ECG) Findings
Description: Abnormal ECG findings included are high and low Heart Rate (HRT), high and low PQ/PR interval (PQ/PR), high and low QRS interval (QRS), high and low QT interval (QT), high and low QTCB interval (QTcB), high and low QTcF interval (QTcF), high and low RR interval (RR), high and low T Wave, high and low U Wave, high and low ECG. The 12 Lead ECG was recorded after participants were in a semi-supine position for at least 5 minutes. Only participants with abnormal ECG findings are presented in the table below.
Time Frame: Up to Day 35
Population: as for outcome 9
Measure: Number; unit: participants
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Number analyzed (Participants) | 7 | 9
participants
  HIGH- HRT ECG ; n=7, 9 | 1 | 0
  LOW- HRT ECG; n=7, 9 | 0 | 0
  HIGH- PQ (PR); n=7, 9 | 0 | 1
  LOW- PQ (PR); n=7, 9 | 0 | 0
  HIGH- QRS; n=7, 9 | 0 | 0
  LOW- QRS; n=7, 9 | 0 | 0
  HIGH- QT; n=7, 9 | 0 | 2
  LOW- QT; n=7, 9 | 0 | 0
  HIGH- QTcB; n=5, 8 | 0 | 2
  LOW- QTcB; n=5, 8 | 0 | 0
  HIGH- QTcF; n=5, 8 | 0 | 2
  LOW- QTcF; n=5, 8 | 0 | 0
  HIGH- RR; n=5, 8 | 0 | 0
  LOW- RR; n=5, 8 | 1 | 0
  HIGH- T WAVE; n=7, 9 | 0 | 0
  LOW- T WAVE; n=7, 9 | 0 | 0
  HIGH- U WAVE; n=1, 0 | 0 | 0
  LOW- U WAVE; n=1, 0 | 0 | 0
  HIGH- ECG; n=7, 9 | 0 | 0
  LOW- ECG; n=7, 9 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 35
Description: All participants who received at least 1 dose of study medication (whether or not they were withdrawn prematurely) and had safety follow-up data were included in safety population. .All AE's and SAE's were collected following the first dose, as well as those that started prior to dosing and worsened on or after the first dose.
Arm/Group | Normal Liver Function | Moderate Hepatic Impairment
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/9
Other Adverse Events (participants affected / at risk) | 3/7 | 5/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Liver Function (N=7) | Moderate Hepatic Impairment (N=9)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Normal Liver Function (N=7) | Moderate Hepatic Impairment (N=9)
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 1 | 3
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 3
Oedema Peripheral (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 1
Liver Tenderness (Hepatobiliary disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Micturition Urgency (Renal and urinary disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.